CLINICAL TRIAL: NCT00790985
Title: Phase 3. Efficacy of Flavocoxid Compared With Naproxen in Subjects With Moderate-severe Osteoarthritis (OA) of the Knee
Brief Title: Efficacy of Flavocoxid 500 mg Compared With Naproxen 500 mg in Subjects With Moderate-severe Osteoarthritis of the Knee
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Primus Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LOA-04P
Record Dates: First submitted 2008-01-16; First posted 2008-11-14 (Estimated); Results first posted 2022-11-01 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2015-10

CONDITIONS: Osteoarthritis of Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — flavocoxid; Naproxen

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- flavocoxid 500 mg (Experimental): flavonoid mixture
  Interventions: Dietary Supplement: flavocoxid
- naproxen (Active Comparator): nonsteroidal anti-inflammatory drug
  Interventions: Drug: Naproxen

INTERVENTIONS:
Dietary Supplement: flavocoxid — medical food
  Other Names: Limbrel
  Arms: flavocoxid 500 mg
Drug: Naproxen — antiinflammatory drug
  Other Names: naprosyn
  Arms: naproxen

SUMMARY:
To compare flavocoxid with naproxen for patients with moderate to severe osteoarthritis of the knee.

DETAILED DESCRIPTION:
Efficacy of flavocoxid 500 mg compared with naproxen 500 mg in subjects with moderate-severe osteoarthritis of the knee.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to read and understand informed consent and questionnaires in English.
* Adults of either gender age 35-75 years, in general good health.
* Established X-ray diagnosis of osteoarthritis of at least one knee.
* Taken NSAID including COX-2 (cyclo-oxygenase-2) inhibitor in full therapeutic dose for at least one month prior to screening.
* Able and will to discontinue osteoarthritis medications until flare criteria met.
* BMI</= 45
* Subjects must rate target knee at least 5 out of 10 on discomfort VAS (visual analogue scale) at baseline visit.
* Have an increase of at least 15mm on a 100mm pain VAS (visual analogue scale) from screening to baseline visit.
* Must use acceptable birth control if female.
* Screening fecal occult must be negative.
* Able to attend all required visits
* Physical Therapy is allowed as long as the type and frequency remains unchanged for the duration of the study.

Exclusion Criteria:

* Refusal to sign consent.
* Inability to attend all clinic visits
* Grade 0-1 K-L changes in both knees or grade 4 K-L changes in either knee on standing A/P radiograph
* Pregnant or lactating women
* History of serious cardio-vascular disease.
* Recurrent arrythmias, except paroxysmal tachycardia, cardiomyopathy, myocardial infarct within one year of screening.
* History of chronic esophageal, gastric or duodenal disease
* History of upper GI bleeding within the past 2 years.
* Any GI disorder associated with malabsorption
* Any musculo-skeletal or neurological condition that results in pain or gait disturbance that might confound evaluation of target knee.
* Uncontrolled Diabetes Mellitus
* History of bleeding disorder or concurrent use of coumadin or any agent used to reduce blood clotting or platelet adhesiveness.
* Concurrent use of any anti-arthritic medication, including corticosteroids regardless of the reason for use. (low dose aspirin for cardioprotection is allowed)
* History of chronic renal disease with creatinine >2.0 or nephrotic syndrome with 24 hour protein excretion >1000mg.
* Intra-articular injection of any hyaluronic acid preparation in the target knee joint within 4 months of baseline visit.
* Intra-articular injection of a corticosteroid in the target knee joint within 2 months of the baseline visit.
* BMI>45
* History of allergic reaction to flavonoid or flavan containing foods or products (example: red wine, colored fruits and vegetable, brazil nuts, tea, natto)
* History of allergy to aspirin, naproxen or other NSAID
* History of substance abuse including alcohol, or any psychiatric condition that may impair the subject's ability to comply with the study requirements.
* Any medical condition that, in the opinion of the investigator, might put the subject at undue risk or might interfere with the subject's ability to participate in the study.
* Participation in another clinical trial within 30 days or 7 half lives of the study agent, whichever is longer, of the screening visit.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2008-01; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul H Caldron, DO, FACP, Study Director — AmeRuss Clinical Trials LLC, USA

IPD SHARING:
Plan to Share IPD: No
interested researchers may contact sponsor

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects presented to their providers medical clinic At Screening anti-inflammatory meds discontinued. At Baseline inclusion, exclusion measured At Baseline randomization for eligible participants
Groups:
- Naproxen 500 mg: nonsteroidal anti-inflammatory drug
  Naproxen: antiinflammatory drug
Period: Overall Study
Arm/Group | Flavocoxid 500 mg | Naproxen 500 mg
Started | 108 | 115
Completed | 106 | 114
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Flavocoxid 500 mg | Naproxen 500 mg | Total
Number analyzed (Participants) | 108 | 115 | 223
Age, Categorical [Count of Participants; unit: Participants] — Population: 2 randomized to intervention discontinued prior to completion
  1 randomized to placebo discontinued prior to completion
  Participants
    number analyzed (Participants) | 106 | 114 | 220
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 100 | 105 | 205
    >=65 years | 6 | 9 | 15
Age, Continuous [Mean (Inter-Quartile Range); unit: years] — Population: 2 randomized to intervention discontinued prior to completion
  1 randomized to placebo discontinued prior to completion
  years
    number analyzed (Participants) | 106 | 114 | 220
    (all) | 60.64 [53 to 69] | 61.08 [54 to 68] | 60.86 [53 to 69]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 2 randomized to intervention discontinued prior to completion
  1 randomized to placebo discontinued prior to completion
  Participants
    number analyzed (Participants) | 106 | 114 | 220
    Female | 93 | 90 | 183
    Male | 13 | 24 | 37
Region of Enrollment [Count of Participants; unit: Participants] — Population: 2 randomized to intervention discontinued prior to completion
  1 randomized to placebo discontinued prior to completion
  Participants
    United States: number analyzed (Participants) | 106 | 114 | 220
    United States | 106 | 114 | 220

OUTCOME MEASURES:

1. Primary Outcome: Western Ontario and McMaster Universities Arthritis (WOMAC) Composite Score: Percent Change From Baseline to Week 12.
Description: WOMAC is a composite of subscales: pain - 5 questions, stiffness - 2 questions, physical function - 17 questions. Subject answers each question as none=0, slight=1, moderate=2, very=3 and extreme=4 of pain, stiffness and difficulty of function. Scores for each subscale are summed, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function. Individual question scores are then summed to form a raw score ranging from 0 (worst) to 96 (best). Raw scores are normalized by multiplying each score by 100/96. This produces a reported WOMAC Score of between 0 (worst) to 100 (best).The higher the score of the units on the scale, the better the outcome.
  For each individual subject, the percent change from baseline to Week 12 in the WOMAC composite score is calculated as 100 x (week 12 minus baseline)/baseline. The higher the percent change, the better the outcome. The percent changes from baseline to Week 12 are then compared between Flavocoxid and Naproxen.
Time Frame: As measured at Baseline and Week 12
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Naproxen | Flavocoxid 500 mg
Number analyzed (Participants) | 106 | 114
percentage of change | 85.75 (9.83) | 69.97 (7.34)

ADVERSE EVENTS:
Time Frame: Screening to Week 12
Groups:
- Flavocoxid 500 mg: Intervention started at Baseline 500 mg BID (two times daily)
- Naproxen 500 mg: Comparator started at Baseline 500 mg BID (two times daily)
Arm/Group | Flavocoxid 500 mg | Naproxen 500 mg
All-Cause Mortality (participants affected / at risk) | 0/108 | 0/115
Serious Adverse Events (participants affected / at risk) | 0/108 | 0/115
Other Adverse Events (participants affected / at risk) | 21/108 | 39/115
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Flavocoxid 500 mg (N=108) | Naproxen 500 mg (N=115)
nausea dyspepsia (Gastrointestinal disorders) | 21 (21) | 39 (39)
edema (Vascular disorders) | 2 (2) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days